CLINICAL TRIAL: NCT00803491
Title: Health Related Quality of Life After a Self-promoting Problem-based Learning Program for People With Rheumatic Diseases: a Randomized Controlled Trial
Brief Title: Health Related Quality of Life After a Self-promoting Learning Program for People With Rheumatic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spenshult Hospital (Other)
Collaborators: The Swedish Rheumatism Ass (Other); County Council of Halland, Sweden (Other Government)
Responsible Party: Stefan Bergman, Research Director, R&D-centre Spenshult Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FOUS08001
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Rheumatic Diseases
Keywords: Rheumatic diseases; Problem based learning; Health-related quality of life; Empowerment; Self-care
MeSH Terms: conditions — Rheumatic Diseases; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Problem based learning program (Experimental): PBL intervention - a self-promoting PBL program for patients with rheumatic diseases.
  Interventions: Other: Problem based learning
- Control group (Active Comparator): Traditional rheumatological care.
  Interventions: Other: Traditional rheumatology care.

INTERVENTIONS:
Other: Problem based learning — Group sessions under supervision from a nurse. Each group including 8 subjects. 10 occasions during a period of one year.
  Arms: Problem based learning program
Other: Traditional rheumatology care. — Individually base.
  Arms: Control group

SUMMARY:
Randomized controlled trial including 200 subjects with rheumatic diseases. Subjects will be randomized to either a self-promoting problem based learning (PBL) program or a control group with traditional care. The hypothesis is that a PBL program will improve health-related quality of life, empowerment and self-care ability.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have one or several rheumatic diseases diagnosed more than a year.
* Subjects should have musculoskeletal pain, sleep disturbances and fatigue, overwhelming number of days during the last three months.
* Subjects should be registered on the waiting list to the rheumatologic clinic.

Exclusion Criteria:

* Subjects with difficulties speaking and/or read Swedish.
* Subjects with difficulties travelling to the clinic.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life as measured by SF-36 | Baseline, after intervention and six, twelve and thirtysix months after

SECONDARY OUTCOMES:
Empowerment as measured by ASES-S | Baseline, after intervention and six, twelve and thirtysix months after
Empowerment measured by SWE-RES-23. | Baseline, after intervention and six, twelve and thirtysix months after
Self-care ability measured by ASA-A. | Baseline, after intervention and six, twelve and thirtysix months after
Sense of coherence (SOC). | Baseline, after intervention and six, twelve and thirtysix months after

CONTACTS AND LOCATIONS:
Overall Officials: Susann Arvidsson, PhD-student, Principal Investigator — R&D-centre Spenshult; Stefan Bergman, MD, PhD, Study Director — R&D-centre Spenshult; Barbro Arvidsson, Professor, Study Chair — R&D-centre Spenshult; Bengt Fridlund, Professor, Study Chair — University of Jönköping, Sweden; Pia Tingström, PhD, Study Chair — University of Linköping
Locations (1):
- Spenshult Hospital, Oskarström, Sweden